CLINICAL TRIAL: NCT03788811
Title: Assessment of ERG Components to Discriminate Between Schizophrenia and Bipolar Disorder Type I
Brief Title: ERG Components in Schizophrenia and Bipolar Disorder Type I
Status: Active, not recruiting | Type: Observational
Sponsor: diaMentis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: dM/CL-01
Record Dates: First submitted 2018-12-20; First posted 2018-12-28 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia; Bipolar I Disorder
Keywords: Retinal Signal; Schizophrenia; Bipolar I Disorder; Support to diagnostic; ERG; Mental Disorder
MeSH Terms: conditions — Schizophrenia; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Control subjects: Control subjects who do not have a lifetime diagnosis of SZ, BP, other psychotic disorder, recurrent mood disorder or have not met criteria for a major depression episode in the last 12 months according to DSM-V criteria.
  Interventions: Device: ERG assessment (RSPA)
- Patients with schizophrenia (SZ): Patient with a diagnosis of schizophrenia for at least 12 months, that resulted in a diagnosis with a Structured Clinical Interview for DSM-5 (SCID-5-CT).
  Interventions: Device: ERG assessment (RSPA)
- Patients with bipolar disorder Type I (BP1): Patient with a diagnosis of bipolar disorder Type 1 for at least 12 months, that resulted in a diagnosis with a Structured Clinical Interview for DSM-5 (SCID-5-CT).
  Interventions: Device: ERG assessment (RSPA)

INTERVENTIONS:
Device: ERG assessment (RSPA) — Processing and analysis of retinal signals

SUMMARY:
This study will further assess ERG components obtained with different ERG devices, to be considered in a prediction model for each diagnosis. The prediction models are diaMentis proprietary software used as an ERG-based diagnostic test (classified as a Software as Medical Device, SaMD) to support the diagnosis of schizophrenia and bipolar disorder type I. They involve the processing and analysis of specific retinal biosignatures (RSPA) with the support of statistical and mathematical modelling processes e.g. machine learning and statistical learning.

DETAILED DESCRIPTION:
The technology under development by diaMentis is defined as a Software as a Medical Device (SaMD); it will be used in combination with an electroretinogram (ERG). This study will be performed using three different ERG devices, currently marketed and cleared by the health authorities (Espion, UTAS and RETeval) to support the analytical, scientific and performance validity of the SaMD.

Anomalies detected by ERG provide an objective measure that may reflect specific underlying dysfunctions in patients and thus hold promise to confirm relevant biosignatures in psychiatric disorders. Significant differences between patients with SZ, BPI and control subjects have been found despite confounding factors; this trial is required to better define the impact of patient characteristics on ERG features with a potential to refine the interpretation of results.

This is a multicenter study. Three hundred subjects will be enrolled into three groups: 100 SZ patients, 100 BPI patients and 100 control subjects (healthy volunteers).

The primary objective is to further characterize the ERG components in SZ and BPI patients in order to develop prediction models that discriminate each pathology.

The secondary objectives are the evaluation of the repeatability and reproducibility of the analysis of the ERG components in control subjects, the assessment of the reliability of ERG prediction score for patients following a repeat test, and the evaluation of the impact of different ERG devices on the data generated and the prediction models.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent;
* 18 to 50 years old;
* Patient with a likely diagnosis of SZ or BPI for at least 12 months, that resulted in a diagnosis of SZ or BPI with a Structured Clinical Interview for DSM-5 (SCID-5-CT);
* Control subjects who do not have a lifetime diagnosis of SZ, BP, other psychotic disorder, recurrent mood disorder or have not met criteria for a major depression episode in the last 12 months according to DSM-V criteria.

Exclusion Criteria:

* Control subjects taking antipsychotic drugs (other prescription medicines are allowed);
* Control subjects with a first-degree relative with SZ, BP, other psychotic disorder or recurrent major depressive disorder;
* Patient currently in an acute inpatient unit and not stable (i.e. experiencing an acute exacerbation of psychosis or mania);
* Diagnosed dementia, Parkinson's disease, autism or other pervasive developmental disorders or seizure disorders (such as epilepsy);
* Substance use disorder within the last 6 months;
* Any known diagnosis of ophthalmological abnormalities, such as diabetic retinopathy, glaucoma, change in intraocular pressure, macular degeneration, other retinal pathologies, congenital color vision deficiencies, strabismus or cataract;
* Any person contra-indicated for an ERG test, including active corneal or conjunctival disease (e.g. pink eye or conjunctivitis), infection or a ruptured globe;
* Subjects in recovery phase following cataract surgery or post LASIK refractive surgery or trabeculectomy or any surgical/laser intervention, suspected penetrating ocular injury, ocular prosthesis or severe photophobia;
* Any person unable to or unwilling to participate in a psychiatric evaluation or ERG testing, including, in the clinical judgment of the Principal investigator, subjects with cognitive impairment that compromises their ability to participate meaningfully in a SCID-5-CT interview.
* Any subject during the course of the study that is pregnant or intends on becoming pregnant and/or receives or intends to receive fertility treatments. Subjects becoming pregnant during study will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patient with a likely diagnosis of SZ or BPI for at least 12 months, that resulted in a diagnosis of SZ or BPI with a Structured Clinical Interview for DSM-5 (SCID-5-CT); and control subjects who do not have a lifetime diagnosis of SZ, BP, other psychotic disorder, recurrent mood disorder or have not met criteria for a major depression episode in the last 12 months according to DSM-V criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-07-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in ERG components vs control ERG with full-field ERG stimulation conditions. | Three ERG assessments within 6 weeks.
  ERG components are retinal signal features (signal amplitude vs time) in the electrical signal recorded up to 100 msec post stimulation.
Differences in ERG components vs control ERG with Photopic Negative Response (PhNR) ERG stimulation conditions. | Three ERG assessments within 6 weeks.
  ERG components are retinal signal features (signal amplitude vs time) in the electrical signal recorded up to 250 msec post stimulation.
Differences in ERG components vs control ERG with On-Off ERG stimulation conditions. | Three ERG assessments within 6 weeks.
  ERG components are retinal signal features (signal amplitude vs time) in the electrical signal recorded up to 300 msec post stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Hariton, PhD, DSc, Study Director — diaMentis Inc.
Locations (19):
- United States (11):
  - Collaborative Neuroscience Research LLC, Garden Grove, California
  - Synergy San Diego, Lemon Grove, California
  - Collaborative Neuroscience Research LLC, Torrance, California
  - Segal trials West Broward Outpatient Site, Lauderhill, Florida
  - Segal Trials Miami Lakes Medical Research, Miami Lakes, Florida
  - McLean Hospital, Belmont, Massachusetts
  - Rutgers University Behavioral HealthCare, Piscataway, New Jersey
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - University of Rochester Medical Center, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - University Hills Clinical Research, Irving, Texas
- Australia (3):
  - Monash Medical Centre, Clayton, Victoria
  - Barwon Health University Hospital, Geelong, Victoria
  - Albert Road Clinic, Melbourne, Victoria
- Canada (5):
  - Queen's University, Kingston, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
  - Institut Universitaire en Santé Mentale de Montréal, Montreal, Quebec
  - Douglas Mental Health University Institute, Montreal, Quebec
  - CISSS-CA Hôpital de Saint-Georges, Saint-Georges, Quebec

IPD SHARING:
Plan to Share IPD: No